CLINICAL TRIAL: NCT04685707
Title: Visual Feedback Monitoring During Exercise in Individuals With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-607
Record Dates: First submitted 2020-12-10; First posted 2020-12-28 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFFS, then Control (Experimental): Participants first performed the HFFS (increased hip flexion) exercise session. After a washout period of at least 24h, they then performed the Control (walking/running) exercise session.
  Interventions: Device: Visual feedback monitoring system (HFFS); Other: Control
- Control, then HFFS (Experimental): Participants first performed the Control (walking/running) exercise session. After a washout period of at least 24h, they then performed the HFFS (increased hip flexion) exercise session.
  Interventions: Device: Visual feedback monitoring system (HFFS); Other: Control

INTERVENTIONS:
Device: Visual feedback monitoring system (HFFS) — Participants will follow the exercise monitoring system's instructions displayed on a TV. Treadmill walking speed will be set at a comfortable walking speed.
Other: Control — Participants will monitor the intensity of exercise independently using a standard heart rate monitor and control it by adjusting the treadmill speed (walking speed).

SUMMARY:
Exercise has been shown to offer numerous health benefits and be particularly important in preventing weight gain or regain for people with obesity. Exercise guidelines can be difficult to interpret and apply independently and do not address specific exercise limitations in individuals with obesity. The exercise monitoring system proposed in this study might provide a new method to meet aerobic exercise guidelines independently with reduced risk of injury.

The exercise monitoring system controls, in real-time, the intensity of an exercise session consisting of treadmill walking. During treadmill walking, the exercise monitoring system will instruct participants to increase or decrease how much participants raise their knees and swing their arms while maintaining a smooth contact with the ground, based on real-time readings of the participants' heart rate.

In this clinical trial, each participant will perform a control and an experimental training session. Both training sessions will include four blocks of 7 minutes of treadmill walking alternated with three periods of rest (3 min). In the control session, participants will monitor the intensity of exercise independently using a standard heart rate monitor and control it by adjusting their walking speed. In the experimental session, each participant will follow the exercise monitoring system instructions displayed on a TV, and treadmill walking speed will be set at a comfortable walking speed. Target heart rates of 60% HRR will be used as the exercise intensities in both training sessions. The investigators will examine energy expenditure, heart rate, and kinematic measures under control and experimental conditions. The goals of this clinical trial are to determine the effect of exercising with the exercise monitoring system in individuals with obesity. The investigators hypothesized that the experimental session will result in higher total energy cost and efficiency than the control session; and in lower heart rate error, tibial positive peak accelerations and feedback errors than the control session.

The results of this study will inform proposals for larger interventions that will focus on 1) testing different types of obesity and osteoarthritis, 2) adding a resistance-training component, and 3) integrating a diet intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30.0 kg/m2 and ≤ 40.0 kg/m2
* Age 20 to 45 years;
* Able to understand spoken English at the level needed to:
* understand and follow instructions for equipment setup, testing, and task performance
* answer questions related to effort and preference
* be able to understand consent document and provide informed assent

Exclusion Criteria:

* Any signs or symptoms suggestive of cardiovascular, pulmonary, metabolic, or renal disease.
* Any injury or health condition that affects the ability to walk on a treadmill.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Southern Mississippi, Hattiesburg, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: HFFS Session
Arm/Group | HFFS, Then Control | Control, Then HFFS
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0
Period: Washout
Arm/Group | HFFS, Then Control | Control, Then HFFS
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0
Period: Control Session
Arm/Group | HFFS, Then Control | Control, Then HFFS
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants were randomized to receive all interventions:
  Visual feedback monitoring system (HFFS): Participants will follow the exercise monitoring system's instructions displayed on a TV. Treadmill walking speed will be set at a comfortable walking speed.
  Control: Participants will monitor the intensity of exercise independently using a standard heart rate monitor and control it by adjusting the treadmill speed (walking speed).
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Energy Expenditure (Oxygen Consumption)
Description: Energy expenditure was evaluated from oxygen consumption (ml/kg/min) measured during the exercise and recovery bouts using a breath-by-breath portable metabolic analyzer (K5, COSMED, Rome, Italy).
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: ml/kg/min
Groups:
- HFFS: Visual feedback monitoring system: Participants will follow the exercise monitoring system's instructions displayed on a TV. Treadmill walking speed will be set at a comfortable walking speed.
Arm/Group | HFFS | Control
Number analyzed (Participants) | 20 | 20
ml/kg/min | 20.2 (5.8) | 22.8 (6.1)

2. Primary Outcome: Heart Rate (Bpm)
Description: Average heart rate (bpm) during steady state period of exercise.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | HFFS | Control
Number analyzed (Participants) | 20 | 20
bpm | 149 (4.5) | 151 (3.8)

3. Primary Outcome: Percentage of Strides With Tibia Peak Positive Accelerations Above 3g
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: % of strides
Arm/Group | HFFS | Control
Number analyzed (Participants) | 20 | 20
% of strides | 23.8 (27.6) | 54.0 (31.0)

4. Secondary Outcome: Mean Tibial Positive Peak Acceleration
Description: Tibia axial accelerations were calculated using an IMU (Xsens Technologies BV, Enschede, Netherlands) aligned in the long axis of the participant's tibia attached to the anteromedial aspect of the distal tibia using double-sided adhesive tape. The mean peak positive acceleration (PPA) was calculated as the mean tibia PPA across all recorded strides for both sides during the exercise above 3g.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: g
Arm/Group | HFFS | Control
Number analyzed (Participants) | 20 | 20
g | 3.5 (0.2) | 4.0 (0.9)

5. Secondary Outcome: Heart Rate Error
Description: Heart rate error (HRerr) was calculated as the absolute error between the target heart rate (HRtarget) and the actual heart rate during the steady state exercise. HRtarget corresponded to 60% heart rate reserve (HRR) of each participant. HRR was calculated as the difference between the estimated maximal heart rate and the resting heart rate. Maximal heart rate was estimated using the 220-age formula, and resting heart rate was measured using the heart rate monitor after at least 4 min of seated rest at the beginning of each session.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | HFFS | Control
Number analyzed (Participants) | 20 | 20
bpm | 3.3 (2.0) | 2.8 (1.5)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | HFFS | Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT04685707/Prot_SAP_000.pdf